CLINICAL TRIAL: NCT05998343
Title: Improving Social Isolation and Loneliness in Older Adults Discharged From the Emergency Department - Comparing an Intergenerational Versus Same Generation Peer-support Intervention Versus Common Wait List Control Group in a Three Arm RCT
Brief Title: Intergenerational Program for Social Isolation and Loneliness in Older Adults Discharged From the Emergency Department
Acronym: SIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: North York General Hospital (Other); Sunnybrook Research Institute (Other); University of Toronto (Other); Bolton Clarke Research Institute (Unknown); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-0074-E
Record Dates: First submitted 2023-07-24; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Social Isolation; Loneliness; Geriatric
Keywords: Loneliness; Social Isolation; Emergency Department; Geriatrics; Geriatric Psychiatry; Family Medicine; Randomized Clinical Trial
MeSH Terms: conditions — Social Isolation; Emergencies

STUDY DESIGN:
Intervention Model Description: This study is a three-arm outcome assessor blinded randomized controlled trial will follow SPIRIT reporting guidelines and is part of a program of research that adheres to the ORBIT model for developing complex behavioural interventions.
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes will be assessed after 12 weeks by a research assistant who is blinded to the intervention group and who has had no prior contact with the participants. Participants will also be instructed not to reveal the intervention they have received to any research staff.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HOW R U? intervention delivered by same-generation peer volunteer (Experimental): HOW R U?
  Interventions: Behavioral: Same-Generation Peer Support HOW R U?
- HOW R U? intervention delivered by intergenerational volunteer (Experimental)
  Interventions: Behavioral: Intergenerational HOW R U?
- Waitlist control group (No Intervention): After the primary outcome assessment at 12 weeks, control group participants will be offered HOW R U? intervention support outside of the main trial. They will be allowed to choose either intergenerational or same-generation versions.

INTERVENTIONS:
Behavioral: Intergenerational HOW R U? — 1-on-1 discussion over telephone with a trained volunteer aged 19-39 years old who has received training to provide strength-based support sessions weekly for 12 weeks.
  Arms: HOW R U? intervention delivered by intergenerational volunteer
Behavioral: Same-Generation Peer Support HOW R U? — 1-on-1 discussion over telephone with a trained volunteer aged 60 years or older who has received training to provide strength-based support sessions weekly for 12 weeks.
  Arms: HOW R U? intervention delivered by same-generation peer volunteer

SUMMARY:
Social isolation and loneliness worsens older adults' risk of dementia, quality of life, and death as much as smoking. Older adults are more likely to use emergency services and are also more likely to experience social isolation and loneliness than younger people. The emergency department is a new setting to screen for social isolation and loneliness in older adults and help accordingly.

Social isolation and loneliness are experienced differently by different older adults. Different interventions combatting social isolation and loneliness may work better for different people, and little is known about older adult's preferences for specific types of interventions.

HOW R U? is an effective and feasible intervention using same-generation peer support offered by trained hospital volunteers to reduce social isolation and loneliness in older adults. In partnership with the Australian developer of HOW R U?, this study will compare an intergenerational HOW R U? intervention using younger volunteers with the same-generation peer support intervention and a waitlist control arm.

The investigators partnered with the staff of emergency departments and family medicine clinics to identify people who will benefit from an intervention combatting, and Volunteer Services to recruit volunteers.

The investigators hypothesize that the older adults who receive the intergenerational HOW R U? intervention will have a greater improvement in social isolation and loneliness.

DETAILED DESCRIPTION:
Introduction:

Social isolation and loneliness (SIL) worsens mortality and other outcomes among older adults as much as smoking. The investigators previously tested the impact of the HOW R U? intervention using peer support from similar aged volunteers and demonstrated reduced SIL among older adults discharged from the Emergency Department (ED). Generativity, defined as "the interest in establishing and guiding the next generation" can provide an alternative theoretical basis for reducing SIL via intergenerational programs between members of younger and older generations. The current study will examine the impact of younger intergenerational volunteers providing the HOW R U? intervention. As part of a program of research following the Obesity-Related Behavioral Intervention Trials (ORBIT ) model, findings of this RCT will be used to define which intervention characteristics are most effective in reducing SIL. This trial builds on feasibility work conducted in the investigators' previous trial (NCT 05228782).

Methods and Analysis:

The investigators will compare the use of the same-generation peer support HOW RU? intervention to support by intergenerational volunteers. The investigators will use a common wait list control group in this three-arm randomized controlled trial (RCT).

Trained volunteers will deliver 12 weekly telephone support calls. The investigators will recruit 141 participants ≥70 years of age with baseline loneliness (six-item De Jong loneliness score of 2 or greater) from two EDs. Research staff will assess change in loneliness (De Jong Loneliness Scale), social isolation (Lubben's Social Network Scale), depression (Geriatric Depression Score), quality of life (EQ-5D-5L), functional status (Older Americans Resource Scale), generativity (Loyola Generativity Scale), and perceived benefit at baseline (subjective Likert scale), at 12-14 weeks, and 24-26 weeks post-intervention. The study will follow the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines.

Ethics and Dissemination:

The participating research ethics boards have granted ethics approval, and the participants randomized to the waitlist control group will be offered their choice of intergenerational or same-generation HOW R U? interventions after 12 weeks. Results will be shared through journal publications, conference presentations, social media, and through the International Federation of Emergency Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Any community-dwelling person 70 years of age and older receiving care from the ED, Family Medicine, or Geriatric clinics at the two participating sites (MSH and NYGH) will be eligible.
* Baseline de Jong loneliness scores of 2.0 will be required for participation in the trial.

Exclusion Criteria:

* Age less than 70 years;
* Patients with communication problems (critically ill, unconscious, language barrier, speech impairment or otherwise unable to provide consent), or admission to a hospital for > 72 hours.
* Patients with severe cognitive impairment or those living in nursing homes who are dependent on others for their activity of daily living will be excluded.
* Patients without any mobile phone or landline.

Volunteers:

* Volunteers will be 60 years of age or older to qualify as peer-support volunteers.
* Volunteers will be 19-39 years of age to qualify as intergenerational volunteers.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in loneliness using De Jong Gierveld 6-item Loneliness Scale from Baseline to 12 Weeks | Measure at baseline, at 12 weeks (primary outcome) and 24 weeks (sustainability)
  The minimum value is 0 and the maximum value is 6, with the higher value corresponding with a greater degree of loneliness. It is divided into 4 clinically relevant categories: 0-1 = no loneliness, 2-3 = low levels of loneliness, 4-5 = moderate to severe loneliness, and 6 = severe loneliness.

SECONDARY OUTCOMES:
Change in perceived social support using Lubben Social Network Scale | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  The Lubben Social Network Scale is a measure of perceived social support received from the family and friends and consists of 6 items each of which is scored from 0 to 5: none = 0, one = 1, two = 2, three or four = 3, five through eight = 4, nine or more = 5. The total score ranges from 0 to 30, and a score of 12 and lower indicates a status of "at-risk" for social isolation
Change in mood using Geriatric Depression Scale | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  The Geriatric Depression Scale is a 15-item scale of mood that is extensively validated in older populations to screen for depression. Scores range from 0 to 15. A score of 0-4 is considered normal, and a score of 5 or higher is considered indicative of depression with higher scores indicating higher severity of depression.
Change in Quality of Life using Euro-Qual 5 Dimensions 5 Levels | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  EQ-5D-5Lin 5 dimensions. In each dimension, quality of life can be measured from 1 (best quality of life) to 5 (worst quality of life), giving a possible score of 5-25. A higher score indicates worse quality of life. (Euro-Qual 5 Dimensions 5 Levels) scale assesses quality of life
Change in Functional Status using Older Americans Resource Scale | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  The Older Americans Resource Scale (OARS) consists of 7 activities of daily living (ADL) questions and 7 instrumental activities of daily living (IADL) all rated as "without any help" (2 points), "with some help" (1 point), or "completely unable" (0 points). The ADL and IADL scores can be used separately or combined to produce an overall OARS score from 0-28.
Change in self-perceptions of generativity using Loyola Generativity Scale | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  The Loyola Generativity Scale is a 20-item scale with each question answered 0 = statement never applies to you, 1 = statement only occasionally or seldom applies to you, 2 = statement applies to you fairly often, or 3 = statement applies to you very often or nearly always.
  The higher the score, the greater the sense of generativity.
Perceived benefit to participant at 12 weeks | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  Perceived benefit by the participant pre- and post-intervention will be assessed using the question "Compared to working with a volunteer around the same age as you, you think that working with a younger volunteer is:" followed by a 5-point Likert scale with the following options: A lot less helpful for me, a little less helpful for me, about the same for me, a little more helpful for me, or a lot more helpful for me.
Perceived benefit to volunteer at 12 weeks | Measure at baseline, at 12 weeks and 24 weeks (sustainability)
  Perceived benefit by the participant for the volunteer pre- and post-intervention will be assessed using the question "Compared to working with a volunteer around the same age as you, you think that working with a younger volunteer is:" followed by a 5-point Likert scale with the following options: A lot less helpful for the volunteer, a little less helpful for the volunteer, about the same for the volunteer, a little more helpful for the volunteer, or a lot more helpful for volunteer.

OTHER OUTCOMES:
Feasibility and Process Outcome 1 - Participant preference | Measure at 12 weeks
  To assess for participant preference for same-generation peer support versus intergenerational HOW R U? intervention, we will use a 5-point Likert scale with the following options: "I strongly prefer peer support", "I prefer peer support", "neutral", "I prefer intergenerational" and "I strongly prefer intergenerational".

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual level data that support the findings of this study will be available on reasonable request from the Principal Investigator Dr. Jacques Lee (Jacques.lee@sinaihealth.ca) to improve scientific transparency, verify the study findings and generating new knowledge. As this research was supported by public funding, request for commercial purposes will require approval of the funding agency.
Time Frame: 18 months from study completion

REFERENCES:
- [Derived] Zheng D, Rose L, Borgundvaag B, McLeod SL, Melady D, Mohindra R, Sinha S, Wesson V, Wiesenfeld L, Kolker S, Kiss A, Lowthian JA, Lee JS. Impact of an intergenerational program to improve loneliness and social isolation in older adults initiated at the time of emergency department discharge: study protocol for a three-arm randomized clinical trial. Trials. 2024 Jun 28;25(1):425. doi: 10.1186/s13063-024-08250-2. PMID 38943176